CLINICAL TRIAL: NCT00096226
Title: A Phase II Trial Of Neoadjuvant Therapy With Concurrent Chemotherapy And High Dose Radiotherapy Followed By Surgical Resection And Consolidative Therapy For Locally Advanced Non-Small Cell Lung Carcinoma
Brief Title: Paclitaxel, Carboplatin, and Radiation Therapy in Treating Patients Who Are Undergoing Surgery for Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0229; CDR0000389508
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemoradiation, Surgery, Chemotherapy (Experimental): Induction paclitaxel(50 mg/m2 I.V. in a one-hour infusion) and induction carboplatin (AUC 2.0 I.V. in a thirty-minute infusion): 1x/week for 6 weeks. Concurrent radiation therapy (RT): 1.8 Gy/day, 5 fx/week, for a total of 50.4 Gy in 28 fractions plus a boost of 1.8 Gy/day, 5 fx/week, for a total of 10.8 Gy in 6 fractions. Followed by an assessment to determine whether patient will undergo a resection or not. Followed by consolidation paclitaxel (200 mg/m2 I.V. over three hours) and consolidation carboplatin (AUC 6.0 over one hour) q 21 days x 2.
  Interventions: Drug: Induction Carboplatin; Drug: Induction Paclitaxel; Procedure: Resection; Drug: Consolidation Carboplatin; Radiation: Radiation Therapy; Drug: Consolidation Paclitaxel

INTERVENTIONS:
Drug: Induction Carboplatin
Drug: Induction Paclitaxel
Procedure: Resection
Drug: Consolidation Carboplatin
Radiation: Radiation Therapy
Drug: Consolidation Paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving paclitaxel and carboplatin together with radiation therapy before surgery may shrink the tumor so that it can be removed. Giving chemotherapy after surgery may kill any tumor cells remaining after surgery.

PURPOSE: This phase II trial is studying how well giving paclitaxel and carboplatin together with radiation therapy works in treating patients who are undergoing surgery for stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the mediastinal node clearance rate in patients with stage IIIA or IIIB non-small cell lung cancer treated with neoadjuvant induction chemoradiotherapy comprising paclitaxel, carboplatin, and high-dose radiotherapy followed by surgical resection for patients found to be resectable and consolidative chemotherapy comprising paclitaxel and carboplatin.
* Determine the rate of complete pathological response in patients treated with this regimen.
* Determine the feasibility of surgical resection after neoadjuvant induction chemoradiotherapy in these patients.
* Determine disease-free and overall survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Stage IIIA (T1-3 N2) or Stage IIIB (N3, excluding supraclavicular involvement) non-small cell lung cancer documented by biopsy or cytology (Pancoast tumors are eligible if pathologic evidence of mediastinal nodal disease is present);
2. Disease must be measurable;
3. Mediastinal lymph nodes must be proven positive by pathologic review. All patients must undergo mediastinoscopy, thoracoscopy, Chamberlain procedure, or transbronchial needle aspirate to evaluate extent of nodal involvement. Any lymph node assessed by mediastinoscopy and found to be positive will be defined as N2 disease;
4. Patients ≥ 18 years of age;
5. Life expectancy ≥ 6 months;
6. Zubrod performance status 0- 1 (See Appendix II);
7. Pretreatment laboratory values must be as follows: White blood cell count (WBC) count: ≥ 3,000/mm^3; Absolute granulocyte count: ≥ 1,500/mm^3; Platelets: ≥ 100,000/mm3; Total bilirubin: ≤ 1.5 x institutional upper limit of normal (ULN); Serum creatinine: ≤ 1.5 x institutional ULN; Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x institutional ULN; serum albumin: ≥ 3.0 g/dL
8. Baseline forced expiratory volume (FEV1) must be at least 2.0 liters; if less than 2.0 then V/Q scan is required and projected post-operative FEV1 must be > 800 cc based on the following formula using the quantitative Ventilation/perfusion (V/Q) scan: FEV1 = FEV1 x % perfusion to uninvolved lung from quantitative lung V/Q scan report.
9. Patient evaluation and acceptance by thoracic surgery, medical oncology, and radiation oncology; patient must be a potential surgical candidate prior to the initiation of therapy;
10. Women of childbearing potential and male participants must practice an effective method of contraception during the study;
11. Pretreatment evaluations required for eligibility include:

    * A complete medical history & physical examination to include Zubrod performance status, neurologic assessment, recent weight loss, usual weight, concurrent non-malignant disease and therapy;
    * Location, type, and size of measurable lesion must be recorded prior to treatment;
    * Complete blood count (CBC) with differential, platelet count, electrolytes, and Mg++ within 14 days prior to study entry;
    * Twelve-channel serum multiple analysis (SMA-12): Total protein, Albumin, Calcium, Glucose, Blood urea nitrogen (BUN), Creatinine, Alkaline Phosphatase, Lactate dehydrogenase (LDH), Total Bilirubin, serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) within 14 days prior to study entry;
    * Women of childbearing potential must have a negative pre-study serum or urine pregnancy test within 14 days prior to study entry.
    * Mediastinoscopy, thoracoscopy, Chamberlain procedure, or bronchoscopy with transbronchial needle aspirate to evaluate the extent of lymph node involvement;
    * Computed tomography (CT) scan of the chest to include liver, and adrenal glands within 6 weeks prior to study entry;
    * Positron emission tomography (PET) scan within 8 weeks prior to study entry. Any suspicious areas outside of the local regional disease requires documented evaluation of these findings to exclude metastatic disease;
    * CT scan or magnetic resonance imaging (MRI) of the brain within 6 weeks prior to study entry;
    * Electrocardiogram (EKG) and pulmonary function tests including forced vital capacity (FVC), FEV-1, and diffusing capacity of carbon monoxide (DLCO), within 8 weeks prior to study entry; V/Q scan, if applicable, within 8 weeks prior to study entry.
12. Patients must sign a study-specific informed consent prior to study entry.

Exclusion Criteria:

1. Small cell lung cancer; distant metastatic disease;
2. Evidence of clinical or radiographic supraclavicular lymph node involvement;
3. Bronchioalveolar carcinoma with lobar or multilobar involvement;
4. Unintentional weight loss > 5% within 6 months prior to study entry, or Zubrod performance status 2 or greater;
5. Primary tumor location prevents delivery of 60 Gy and simultaneously limiting spinal cord dose to 48 Gy;
6. Patients with malignant pleural effusion;
7. Clinically evident superior vena cava syndrome;
8. Prior systemic chemotherapy or radiation therapy to the thorax;
9. Patients with known hypersensitivity to Cremophor EL;
10. Patients receiving other investigational therapy;
11. Pregnant or lactating women are ineligible, as treatment involves unforeseeable risks to the participant and to the embryo or fetus;
12. Patients with an active serious infection or other serious underlying medical condition that would impair their ability to complete protocol treatment;
13. Dementia or significantly altered mental status that would prohibit the understanding and/or giving of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-09; Primary Completion 2012-04 (Actual); Study Completion 2016-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Suntharalingam, MD, Principal Investigator — University of Maryland Greenebaum Cancer Center
Locations (22):
- United States (22):
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Virginia G. Piper Cancer Center at Scottsdale Healthcare - Shea, Scottsdale, Arizona
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Cancer Institute of New Jersey at Cooper University Hospital - Camden, Camden, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin

REFERENCES:
- [Result] Suntharalingam M, Paulus R, Edelman MJ, Krasna M, Burrows W, Gore E, Wilson LD, Choy H. Radiation therapy oncology group protocol 02-29: a phase II trial of neoadjuvant therapy with concurrent chemotherapy and full-dose radiation therapy followed by surgical resection and consolidative therapy for locally advanced non-small cell carcinoma of the lung. Int J Radiat Oncol Biol Phys. 2012 Oct 1;84(2):456-63. doi: 10.1016/j.ijrobp.2011.11.069. Epub 2012 Apr 28. PMID 22543206
- [Result] Suntharalingam M, Paulus R, Edelman MJ, et al.: RTOG 0229: A phase II trial of neoadjuvant therapy with concurrent chemotherapy and high-dose radiotherapy (XRT) followed by resection and consolidative therapy for LA-NSCLC. [Abstract] J Clin Oncol 28 (Suppl 15): A-7024, 2010.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemoradiation, Surgery, Chemotherapy
Started | 60
Eligible | 57
Eligible and Underwent Surgery | 37
Completed | 57 (Subjects contributing any data to analysis are considered to have completed the study)
Not Completed | 3
Not completed — Ineligible | 2
Not completed — Protocol treatment not started | 1

BASELINE CHARACTERISTICS:
Population: All eligible patients who started protocol treatment.
Groups:
- Chemoradiation, Surgery, Chemotherapy: Chemoradiation, surgery, chemotherapy
  carboplatin
  paclitaxel
  adjuvant therapy
  conventional surgery
  neoadjuvant therapy
  radiation therapy
Arm/Group | Chemoradiation, Surgery, Chemotherapy
Number analyzed (Participants) | 57
Age, Continuous [Median (Full Range); unit: years] | 59 [41 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Mediastinal Nodal Clearance Rate
Description: If at least 12 of the first 21 evaluable patients and at least 27 of the the first 45 evaluable patients have mediastinal nodal clearance (MNC), then a conclusion of a 70% MNC rate (compared to 50%) is made using Simon's two-stage design with 90% power and 10% type I error.
Time Frame: At completion of concurrent chemotherapy and radiation therapy, up to 14 weeks.
Population: Eligible patients who had adequate pathologic information of mediastinal nodal status.
Measure: Number; unit: participants
Arm/Group | Chemoradiation, Surgery, Chemotherapy
Number analyzed (Participants) | 43
participants | 27

2. Secondary Outcome: Percentage of Patients With Complete Pathological Response After Concurrent Chemotherapy and Radiation Therapy
Description: Complete pathologic response is defined as complete resection achieved and no evidence of viable tumor in the entire resection specimen.
Time Frame: At time of surgery (16-18 weeks)
Population: Eligible patients who underwent surgery
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation, Surgery, Chemotherapy
Number analyzed (Participants) | 37
percentage of participants | 8.1 [1.7 to 21.9]

3. Secondary Outcome: Percentage of Patients With Major Surgical Morbidities Within 30 Days of Surgery
Description: The surgical morbidities occurring within 30 days following resection were assessed and graded using the NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0. A major morbidity is considered a grade 3 or higher of any of the following: pneumonitis, infection, atelectasis, chest tube drainage/bronchial stump leak, pneumothorax, chylothorax, cardiac ischemia/infarction, pulmonary thrombosis/embolism, supraventricular atrial arrhythmia, ventricular arrhythmia, post-operative hemorrhage, pulmonary/upper respiratory fistula, pleural effusion, or death.
Time Frame: From 0 to 30 days following surgery (surgery occurs within 16-18 weeks after registration)
Population: Eligible patients who underwent surgery
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation, Surgery, Chemotherapy
Number analyzed (Participants) | 37
percentage of participants | 21.6 [9.8 to 38.2]

4. Secondary Outcome: Percentage of Patients Able to Undergo Surgical Resection
Time Frame: At time of surgery (16-18 weeks)
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation, Surgery, Chemotherapy
Number analyzed (Participants) | 57
percentage of participants | 64.9 [51.1 to 77.1]

5. Secondary Outcome: Distribution of R0, R1, and R2 Resections After Chemotherapy
Description: An R0 resection is defined as a complete resection of all disease with negative margins and the highest lymph node resected negative for residual tumor. An R1 resection is defined as a complete resection of all disease with pathology of positive margins, pathologic evidence of tumor cells in the highest lymph node resected in the mediastinum, or extracapsular nodal spread. An R2 resection is defined as gross residual disease left behind after surgical resection.
Time Frame: At time of surgery (16-18 weeks)
Population: Eligible patients who underwent surgery
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation, Surgery, Chemotherapy
Number analyzed (Participants) | 37
percentage of participants
  R0 | 75.7 [61.9 to 89.5]
  R1 | 24.3 [11.8 to 41.2]
  R2 | 0 [0 to 0]

6. Secondary Outcome: Overall Survival at Two Years
Description: Overall survival time is defined as time from registration to the date of death from any cause. Overall survival rate is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact.
Time Frame: From registration to two years
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation, Surgery, Chemotherapy
Number analyzed (Participants) | 57
percentage of participants | 53.8 [40.0 to 65.8]

7. Secondary Outcome: Progression-free Survival at Two Years
Description: Progression is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions. An event for progression-free survival is the first occurrence of progression or death due to any cause. Progression-free survival time is defined as the time from study entry to the the date progression or death, or last known follow-up (censored) if neither progression nor death occurred. Progression-free survival rate is estimated using the Kaplan-Meier method.
Time Frame: From registration to two years
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation, Surgery, Chemotherapy
Number analyzed (Participants) | 57
percentage of participants | 32.7 [20.9 to 45.0]

8. Secondary Outcome: Distribution of Highest Grade Adverse Event
Description: The number of patients whose highest grade adverse event (AE) reported was 3, 4, or 5 was calculated. Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to AE. Number of patients with highest grade of 3, 4, and 5 are presented.
Time Frame: From start of treatment to end of follow-up, a maximum of 64.3 months
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation, Surgery, Chemotherapy
Number analyzed (Participants) | 57
percentage of participants
  Grade 3 | 49.1 [35.6 to 62.7]
  Grade 4 | 19.3 [10.1 to 31.9]
  Grade 5 | 1.8 [0.0 to 9.4]

ADVERSE EVENTS:
Description: Eligible patients are included. Patients experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Chemoradiation, Surgery, Chemotherapy
Serious Adverse Events (participants affected / at risk) | 19/57
Other Adverse Events (participants affected / at risk) | 57/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemoradiation, Surgery, Chemotherapy (N=57)
Blood/bone marrow - Other (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 3
Arrhythmia NOS (Cardiac disorders) | 1
Myocardial ischemia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Ocular/visual - Other (Eye disorders) | 1
Abdominal distention (Gastrointestinal disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Esophagitis NOS (Gastrointestinal disorders) | 2
Ileus paralytic (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 1
Vomiting NOS (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 1
Fatigue (General disorders) | 2
Pyrexia (General disorders) | 2
Rigors (General disorders) | 1
Hypersensitivity NOS (Immune system disorders) | 1
Serum sickness (Immune system disorders) | 1
Anal infection NOS (Infections and infestations) | 1
Gingival infection (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Wound (Infections and infestations) | 1
Leukopenia NOS (Investigations) | 3
Lymphopenia (Investigations) | 2
Weight decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia NOS (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Headache (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 3
Prolonged chest tube drainage or air leak after pulmonary resection (Respiratory, thoracic and mediastinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hypotension NOS (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemoradiation, Surgery, Chemotherapy (N=57)
Blood/bone marrow - Other (Blood and lymphatic system disorders) | 7
Hemoglobin (Blood and lymphatic system disorders) | 38
Pericardial effusion (Cardiac disorders) | 10
Sinus tachycardia (Cardiac disorders) | 11
Supraventricular arrhythmia NOS (Cardiac disorders) | 10
Vision blurred (Eye disorders) | 3
Constipation (Gastrointestinal disorders) | 25
Diarrhea NOS (Gastrointestinal disorders) | 14
Dry mouth (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 13
Dysphagia (Gastrointestinal disorders) | 33
Esophageal pain (Gastrointestinal disorders) | 10
Esophagitis NOS (Gastrointestinal disorders) | 32
Gastritis NOS (Gastrointestinal disorders) | 3
Mucositis/stomatitis (functional/symptomatic): Esophagus (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 35
Stomatitis (Gastrointestinal disorders) | 5
Vomiting NOS (Gastrointestinal disorders) | 13
Chest pain (General disorders) | 19
Edema: limb (General disorders) | 4
Fatigue (General disorders) | 53
Pain - Other (General disorders) | 11
Pyrexia (General disorders) | 10
Rigors (General disorders) | 4
Hypersensitivity NOS (Immune system disorders) | 7
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 30
Radiation recall syndrome (Injury, poisoning and procedural complications) | 6
Alanine aminotransferase increased (Investigations) | 11
Aspartate aminotransferase increased (Investigations) | 12
Blood alkaline phosphatase increased (Investigations) | 9
Blood bilirubin increased (Investigations) | 5
Blood creatinine increased (Investigations) | 5
Leukopenia NOS (Investigations) | 37
Lymphopenia (Investigations) | 14
Metabolic/laboratory - Other (Investigations) | 6
Neutrophil count (Investigations) | 22
Platelet count decreased (Investigations) | 17
Weight decreased (Investigations) | 26
Anorexia (Metabolism and nutrition disorders) | 34
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 11
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia NOS (Metabolism and nutrition disorders) | 34
Hyperkalemia (Metabolism and nutrition disorders) | 9
Hypermagnesemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 16
Hypocalcemia (Metabolism and nutrition disorders) | 11
Hypokalemia (Metabolism and nutrition disorders) | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 15
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Back pain (Musculoskeletal and connective tissue disorders) | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Chest wall pain (Musculoskeletal and connective tissue disorders) | 17
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Ataxia (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 8
Dysgeusia (Nervous system disorders) | 9
Headache (Nervous system disorders) | 8
Peripheral motor neuropathy (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 28
Anxiety (Psychiatric disorders) | 5
Confusional state (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 12
Pollakiuria (Renal and urinary disorders) | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 10
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 41
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 46
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6
Laryngitis NOS (Respiratory, thoracic and mediastinal disorders) | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 20
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 10
Prolonged chest tube drainage or air leak after pulmonary resection (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 7
Pulmonary/upper respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 5
Rhinitis allergic NOS (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 25
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 6
Dermatology/skin - Other (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 8
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 18
Sweating increased (Skin and subcutaneous tissue disorders) | 7
Hot flushes NOS (Vascular disorders) | 4
Hypotension NOS (Vascular disorders) | 6
Thrombosis (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No